CLINICAL TRIAL: NCT03518307
Title: Epidemiology of Merkel Carcinomas in the Bas-Rhin From 1983 to 2011: General Population Study Based on the Bas-Rhin Cancer Registry
Brief Title: Epidemiology of Merkel Carcinomas in the Bas-Rhin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6840
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Merkel Carcinoma
Keywords: Merkel carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this work is to study demographic, clinical, management (diagnostic and therapeutic) and survival data concerning patients with Merkel's carcinoma in the Lower Rhine, thus obtaining the first French data.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of primary Merkel carcinoma (topographic code C44 morphological code 8247/3)
* Diagnosis made between 1983 and 2011
* Patient residing in the Bas-Rhin at the date of diagnosis
* Patient who has given his consent for the use of his data for research purposes

Exclusion Criteria:

- Refusal to participate in research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients residing in the Bas-Rhin and diagnosed between 1983 and 2011 as having primitive Merkel arcinoma (topographic code C44 morphological code 8247/3)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of demographic, clinical, management (diagnostic and therapeutic) and survival data for patients with Merkel carcinoma in the Lower Rhine region | The period from from January 1st, 1983 to December 31st, 2011 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Dan LIPSKER, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Dermatologie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No